CLINICAL TRIAL: NCT01654081
Title: A Non-randomized Phase II Protocol of Irinotecan for Patients With Previously Treated, Advanced ISG15-positive Non-small Cell Carcinoma of the Lung
Brief Title: A Protocol of Irinotecan for Carcinoma of the Lung
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Susanne Arnold (Other)
Responsible Party: Sponsor-Investigator, Susanne Arnold, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-LUN-90-MCC
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-05

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; POSITIVE NON SMALL CELL CARCINOMA; ISG15; IRINOTECAN
MeSH Terms: conditions — Lung Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Irinotecan (Experimental): Irinotecan 125 mg/m2 on days 1, 8, 15 and 22 of every 6- week cycle
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Irinotecan — Irinotecan 125 mg/m2 on days 1, 8, 15 and 22 of every 6- week cycle

SUMMARY:
The goal of this trial is to demonstrate the potential clinical benefit of irinotecan chemotherapy in patients with a specific NSCLC phenotype, ISG15-positive. The use of irinotecan in subjects with ISG15-positive NSCLC will be associated with an improved rate of clinical benefit (objective response, disease stability, and time to progression) compared to historical controls that were not previously selected for ISG-15 expression.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age or greater with histologically or cytologically confirmed non-small cell lung cancer that is advanced and cannot be treated adequately by radiotherapy or surgery; or metastatic or recurrent disease after at least one prior chemotherapy regimen
* Prior invasive malignancies are allowed, provided at least five years has elapsed since the completion of therapy and enrollment on this protocol.
* All participants must have received at least one prior chemotherapy regimen for metastatic NSCLC; prior adjuvant or neoadjuvant chemotherapy for NSCLC will also be allowed, but will NOT be counted toward the number of regimens for metastatic disease unless patients develop evidence of metastatic disease within six months of the initiation of the adjuvant chemotherapy, indicating resistance to platinum-based therapy. There is no limit on the number of prior regimens allowed, provided the patient meets all other eligibility criteria. Patients who may best benefit from the application of specific targeted therapies (i.e., erlotinib for EGFR exon 19 or 21 activating mutations, or crizotinib for EML4-ALK translocations) will be eligible for this protocol only after documented progression through such targeted therapy AND a platinum-based doublet regimen
* All participants must have the appropriate phenotype on pretreatment screening of tumor tissue or sputa, consisting of ISG15-positive cells by immunohistochemistry (staining score of 4-12, as defined in section 4.2), performed by the UK Department of Pathology, and must agree to have their tissues evaluated for ISG15 expression (a separate informed consent will be requested). Potential participants who have no available tissue for assessment will be offered sputum assessment or tissue biopsy if it can be performed safely, potential disease sites can be safely approached, and only if it is the opinion or their attending physician that participation in this protocol represents their best treatment option at this time. Subjects with assessable material will not be required to undergo a separate biopsy solely for participation in this protocol.
* Subjects must have the following baseline laboratory values (bone marrow, renal, hepatic):
* Adequate bone marrow function:
* Absolute neutrophil count >1000/μL
* Platelet count >100'000/μL
* Serum creatinine < 2.0 mg/dL
* Bilirubin <1.5x normal
* Serum calcium < 12 mg/dl
* Signed Informed Consent
* ECOG Performance Status <2
* Life expectancy > 16 weeks
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >20 mm with conventional techniques or as >10 mm with spiral CT scan, MRI, or calipers by clinical exam. See Section 11 for the evaluation of measurable disease.
* Patients of childbearing potential must be using an effective means of contraception.

The effects of Irinotecan on the developing human fetus are unknown. For this reason and because camptothecins are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of irinotecan administration.

Exclusion Criteria:

* Prior therapy with irinotecan, topotecan, or other camptothecin analog
* Patients whose tumor harbors an EGFR exon 19 or 21 mutation who has not yet received prior therapy with an EGFR-specific tyrosine kinase inhibitor such as erlotinib or gefitinib
* Patients whose tumor harbors an EML4/ALK translocation and who has not yet received crizotinib
* Pregnant or lactating females
* Myocardial infarction or ischemia, or active cerebrovascular disease, within the 6 months before Cycle 1' Day 1
* Uncontrolled clinically significant dysrhythmia
* Prior radiotherapy to an indicator lesion unless there is objective evidence of tumor growth in that lesion
* Uncontrolled metastatic disease of the central nervous system (previously treated, stable disease is allowable on this protocol)
* Radiotherapy within the 2 weeks before registration
* Surgery within the 2 weeks before registration
* Any co morbid condition that' in the view of the attending physician' renders the patient at high risk from treatment complications
* Patients who have had chemotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Patients who are receiving any other investigational agents.
* Patients with known untreated brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Pregnant women are excluded from this study because Irinotecan is a camptothecin with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Irinotecan, breastfeeding should be discontinued if the mother is treated with Irinotecan.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Irinotecan. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Progression-free survival following irinotecan therapy | up to five years after initiation of protocol therapy
  Progression-free survival following irinotecan therapy

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Arnold, M.D., Principal Investigator — Lucille P. Markey Cancer Center at University of Kentucky